CLINICAL TRIAL: NCT04970238
Title: Effect of Levosimendan on Left Ventricular Systolic Function and Heart Failure After PCI in Patients With Acute Anterior Myocardial Infarction-- Multicenter Prospective Randomized Controlled Trial
Brief Title: Effect of Levosimendan on Left Ventricular Systolic Function and Heart Failure After PCI in Patients With Acute Anterior Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zhijun Sun (Other)
Responsible Party: Sponsor-Investigator, Zhijun Sun, Director of the second Department of cardiovascular medicine, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021PS522K
Record Dates: First submitted 2021-06-16; First posted 2021-07-21 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: ST Elevation Myocardial Infarction; Heart Failure
Keywords: Heart Failure; Levosimendan
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Heart Failure | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levosimendan group (Experimental)
  Interventions: Drug: Levosimendan
- placebo group (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Levosimendan — Test drug: drug preparation method: 5ml (12.5mg) levosimendan injection was mixed with 500ml 5% glucose injection, the initial loading dose was 6 µg / kg for 10 minutes, followed by continuous infusion of 0.1 µg/ kg / min for 24 hours.
  Arms: Levosimendan group
Other: placebo — Control drug: 5% glucose injection, intravenous injection method is the same as the experimental group pump dose, the initial load dose of treatment is 6 µg / kg for 10 minutes, followed by continuous infusion of 0.1 µg / kg / min for 24 hours.
  Arms: placebo group

SUMMARY:
Reperfusion therapy for acute ST segment elevation myocardial infarction (STEMI) can significantly reduce mortality, but patients may still have heart failure and adverse cardiovascular events due to massive myocardial loss. About 20% of patients present with acute heart failure (AHF) at admission, It is the most important cause of hospital death in acute myocardial infarction. Because of the large necrotic area of acute anterior myocardial infarction, heart failure still occurs in a considerable number of patients even after revascularization (PCI). Myocardial protection of ischemic myocardium is a hot topic in clinical research.

Both ESC and Chinese heart failure guidelines recommend levosimendan for the treatment of acute decompensated heart failure. A large number of studies have proved that levosimendan can significantly reduce myocardial injury and improve cardiac function in patients with acute STEMI complicated with left ventricular dysfunction and cardiogenic shock compared with placebo. Basic research has confirmed that levosimendan can reduce the myocardial infarction area after acute coronary occlusion, improve the left ventricular function, and exert the effects of anti myocardial ischemia, myocardial injury, myocardial fibrosis, ventricular remodeling and anti apoptosis. However, there is still a lack of early preventive application of levosimendan in acute anterior myocardial infarction after PCI to improve ventricular remodeling and reduce the incidence of heart failure.

The purpose of this study was to investigate the effect of early prophylactic levosimendan on left ventricular remodeling, ischemic myocardial protection and the development of heart failure in patients with acute anterior myocardial infarction after PCI.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old.
* 2. Acute anterior wall myocardial infarction (ECG indicates acute anterior wall, acute anterior wall myocardial infarction, acute extensive anterior wall myocardial infarction).
* 3. The onset time of chest pain was less than 12 hours, and agreed to emergency PCI treatment.
* 4. Be able to understand and sign informed consent voluntarily.

Exclusion Criteria:

* 1. Patients who cannot undergo PCI treatment after coronary angiography, or those who fail to open blood vessels, or refuse to undergo PCI treatment.
* 2. Those whose coronary angiography results indicated myocardial infarction caused by non-coronary artery disease or residual stenosis < 50% after reanalization of myocardial infarction without PCI treatment.
* 3. Patients with old anterior wall myocardial infarction.
* 4. Previous history of cardiac insufficiency.
* 5. Both anterior descending stent implantation, stent restenosis or stent thrombosis.
* 6. Symptomatic hypotension, systolic blood pressure < 90mmHg (still < 90mmHg with IABP)
* 7, body temperature > 38.5℃, or with serious infectious diseases (severe myocarditis, severe pneumonia, severe urinary tract infection, etc.).
* 8. Severe other organ diseases (renal insufficiency: EGFR < 30ml/min, severe liver insufficiency, moderate and severe anemia, malignant tumor, hematologic system diseases, etc.).
* 9. Known or suspected allergy to the active or inactive ingredients of the drug under study.
* 10. Participated in other drug clinical trials within 3 months before the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of heart failure | 6 month
  6 month of heart failure
Major Adverse Cardiovascular Events (MACE) | 6 months
  Mace is defined as cardiovascular death and cardiovascular related readmission
Left ventricular systolic function | 72 hours
  At 72 hours, left ventricular systolic function of AFI is as follows ( PSD, GLS, PSI)

SECONDARY OUTCOMES:
NT-ProBNP | 30 days
  Changes of NT-ProBNP at 72 hours and 30 days
Patient quality of life score | 30 days
  Seattle Angina Questionnaiire is used, The full score of five items in the scale is 100. The higher the score is, the better the condition is.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China